CLINICAL TRIAL: NCT06464523
Title: The Effect of HPV Training on Early Diagnosis Screening and Knowledge Levels of Female Teachers
Brief Title: HPV Education, Early Diagnosis and Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GO 2020/71)
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Female Teachers

STUDY DESIGN:
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face to face education (Experimental): In addition to the standard cervical cancer screening programme service, participants in this group received individual face-to-face health education on HPV and cervical cancer prevention through home visits and were given educational brochures. Participants in this group were interviewed a total of four times (four times face-to-face) during the research process.
  Interventions: Behavioral: Face to face education
- Online education (Experimental): In addition to the standard cervical cancer screening programme service, participants in this group received individual health education on HPV and cervical cancer prevention online via video call via WhatsApp application and were given a digital education brochure. Participants in this group were interviewed a total of four times (four times remotely) during the research process.
  Interventions: Behavioral: Online education
- Control (No Intervention): During the research process, the participants in the control group did not receive any intervention other than the standard cervical cancer screening programme service. During the research process, the participants in the control group were interviewed face-to-face twice. After the termination of the study, health education on protection against HPV and cervical cancer was provided to the volunteer participants by a method they specified and an educational brochure was given.

INTERVENTIONS:
Behavioral: Face to face education — In addition to the standard cervical cancer screening programme service, participants in this group received individual face-to-face health education on HPV and cervical cancer prevention through home visits and were given educational brochures. Participants in this group were interviewed a total of four times (four times face-to-face) during the research period.
  Arms: Face to face education
Behavioral: Online education — In addition to the standard cervical cancer screening programme service, participants in this group received individual health education on HPV and cervical cancer prevention online via video call via WhatsApp application and were given a digital education brochure. Participants in this group were interviewed a total of four times (four times remotely) during the research process.
  Arms: Online education

SUMMARY:
The aim of this study was to determine the effect of health education given to female teachers on HPV knowledge and screening test. The population of the study consisted of all female teachers belonging to the Bucak Directorate of National Education between September 2021 and March 2022. The sample of the study consisted of 144 healthy female teachers who were registered in the institutions affiliated to the District Directorate of National Education between the specified dates, met the inclusion criteria and volunteered to participate in the study. In this study area, with the assumption that the rate of cervical cancer screening test of 70% of the women in the Healthy Life Centre after the trainings would be considered significant, the effect size d=0.18 was calculated to include at least 98 women in 3 groups at 95% power and 0.05 error level. The calculation was performed with the 'G Power 3.1.9.2' package programme. In this context, the total sample of the study was determined as 156 participants, 52 in each group.

ELIGIBILITY:
Inclusion Criteria:

* to volunteer to participate in the study,
* To be between the ages of 30-65,
* being a woman teacher,
* being married
* to be able to make video calls.

Exclusion Criteria:

* being pregnant or in the postnatal period,
* a history of cervical cancer,
* to have hysterectomy operation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Human Papilloma Virus (HPV) Knowledge Scale: | 5-10 minutes
  HPV Knowledge Scale is a knowledge test developed by Waller et al. (2013) to determine the level of knowledge of individuals about HPV agent, HPV screening tests and vaccine. The scale, whose Turkish validity and reliability was conducted by Demir and Özdemir in 2019, has a total of 33 items. The HPV Knowledge Scale consists of four sub-dimensions: general HPV knowledge (items 1-16), HPV screening test knowledge (items 17-22), general HPV vaccine knowledge (items 23-27) and knowledge of the current HPV vaccination programme (items 28-33).

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Bayik Temel A, Daghan S, Kaymakci S, Ozturk Donmez R, Arabaci Z. Effect of structured training programme on the knowledge and behaviors of breast and cervical cancer screening among the female teachers in Turkey. BMC Womens Health. 2017 Dec 7;17(1):123. doi: 10.1186/s12905-017-0478-8. PMID 29216918
- [Result] Kocaoz S, Ozcelik H, Talas MS, Akkaya F, Ozkul F, Kurtulus A, Unlu F. The Effect of Education on the Early Diagnosis of Breast and Cervix Cancer on the Women's Attitudes and Behaviors Regarding Participating in Screening Programs. J Cancer Educ. 2018 Aug;33(4):821-832. doi: 10.1007/s13187-017-1193-8. PMID 28285418
- [Result] Keten HS, Ucer H, Dalgaci AF, Isik O, Ercan O, Guvenc N. Knowledge, Attitude, and Behavior of Teachers Regarding HPV (Human Papillomavirus) and Vaccination. J Cancer Educ. 2021 Jun;36(3):584-590. doi: 10.1007/s13187-019-01668-2. PMID 31840211